CLINICAL TRIAL: NCT04164433
Title: Workplace-based HIV Self-testing (HIVST) and Linkage to Care or Prevention Services Among Men in Private Security Services in Uganda: A Cluster Randomized Trial
Brief Title: Workplace-based HIV Self-testing Among Men in Uganda (WISe-Men)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHSREC 2018-054; HS 2672 (Other: Uganda National Council of Science and Technology)
Record Dates: First submitted 2019-11-09; First posted 2019-11-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections
Keywords: HIV self-testing; Men; Workplace; Security Services; Linkage
MeSH Terms: conditions — HIV Infections; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workplace-based HIV Self-Testing (Experimental): i. Explain the procedure of conducting HIVST & interpret HIV self- test result to the user.
  ii. Demonstrate how to perform the self-test and how to interpret the self-test result.
  iii. Provide appointment card including information on linkage for HIV prevention services and further testing for diagnosis among those with a reactive self-test. Participants with a non-reactive self-test will be referred to HIV prevention services.
  iv. Provide a toll free number for continued consultation
  Interventions: Device: Oral HIV Self-Test (OraQuick)
- Workplace-based standard HIV Testing Services (HTS) (No Intervention): Standard of care following the HIV testing algorithm .

INTERVENTIONS:
Device: Oral HIV Self-Test (OraQuick) — The oral HIV self-test is a device for taking a test which is painless. The user gently swipes the test swab along the upper gums once and the lower gums once. The swab is then inserted inside the test tube provided and results are ready in 20 minutes.
  Arms: Workplace-based HIV Self-Testing

SUMMARY:
This study seeks to determine whether workplace delivery of HIV self-testing will lead to an increase in uptake of HIV testing and subsequent linkage to care or prevention services among men in Uganda.

DETAILED DESCRIPTION:
The current coverage of HIV testing and counseling in Uganda is 60% with only 34% of these being men and only about 55% of males living with HIV know their status (MoH, 2016). The challenges with HIV testing require a new focus and new approaches to reach people with undiagnosed HIV infection.

HIV self-testing (HIVST) is one such innovative approach to making testing more accessible to several under-served populations such as men and key populations (WHO, 2013).

In this regard, this study seeks to determine whether providing HIVST in workplace settings will increase the uptake of HIV testing services among men employed in private security services in Uganda and improve linkage to treatment and prevention services.

Design: Cluster randomized trial in two Ugandan districts

Participants: Male employees of private security companies

ELIGIBILITY:
Eligibility Criteria:

* 18-60 years old
* Employed >6 months in the private security company
* Men who have not tested for HIV before
* Men who tested HIV >one year ago

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 548 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
HIV self-testing | Within one month of the intervention
  Proportion of men who self-report testing after receiving a kit at the workplace

SECONDARY OUTCOMES:
Linkage into HIV care and confirmatory testing following HIV self-testing | measured at 1 and 3 months after intervention
  Proportion of participants who self report confirmatory testing from a health facility for all participants with a reactive-self test
Consistent condom use following HIV self-testing | measured at 1 and 3 months after intervention
  Proportion of participants who use a condom for each sexual encounter in a month.
Initiation of Antiretroviral Therapy (ART) following a confirmatory HIV test | measured at 1 and 3 months after intervention
  Proportion of participants who self report ART initiation following a positive result from a confirmatory HIV test result or evidence of an ART card. Data will be collected using a questionnaire.
Uptake of Voluntary Male Medical Circumcision (VMMC) following HIV self-testing | measured at 1 and 3 months after intervention
  Proportion of previously uncircumcised participants who self report Voluntary Male Medical Circumcision (VMMC).
Uptake of PrEP by Most-At-Risk Populations (MARP) following HIV self-testing | measured at 1 and 3 months after intervention
  Proportion of participants considered as Most-At-Risk Populations (MARP) who initiate Pre-exposure prophylaxis (PrEP)

CONTACTS AND LOCATIONS:
Overall Officials: Patience A. Muwanguzi, Principal Investigator — Makerere University; Nelson K. Sewankambo, Study Director — Makerere University; Noah Kiwanuka, Study Director — Makerere University
Locations (2):
- Uganda (2):
  - Security companies, Hoima
  - Security companies, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muwanguzi PA, Ngabirano TD, Kiwanuka N, Nelson LE, Nasuuna EM, Osingada CP, Nabunya R, Nakanjako D, Sewankambo NK. The Effects of Workplace-Based HIV Self-testing on Uptake of Testing and Linkage to HIV Care or Prevention by Men in Uganda (WISe-Men): Protocol for a Cluster Randomized Trial. JMIR Res Protoc. 2021 Nov 1;10(11):e25099. doi: 10.2196/25099. PMID 34723826
- [Derived] Muwanguzi PA, Kutyabami P, Osingada CP, Nasuuna EM, Kitutu FE, Ngabirano TD, Nankumbi J, Muhindo R, Kabiri L, Namutebi M, Nabunya R, Kiwanuka N, Sewankambo N. Conducting an ongoing HIV clinical trial during the COVID-19 pandemic in Uganda: a qualitative study of research team and participants' experiences and lessons learnt. BMJ Open. 2021 Apr 21;11(4):e048825. doi: 10.1136/bmjopen-2021-048825. PMID 33883157
- See also: The Uganda HIV and AIDS country progress report July 2015-June 2016 — http://www.unaids.org/sites/default/files/country/documents/UGA_2017_countryreport.pdf
- See also: Report on the first international symposium on self-testing for HIV: The legal, ethical, gender, human rights and public health implications of self-testing scale-up — http://apps.who.int/iris/bitstream/handle/10665/85267/9789241505628_eng.pdf;jsessionid=22DEE411C5D604E96F5601F74A42BA89?sequence=1